CLINICAL TRIAL: NCT00332865
Title: Swallow Exercise as Prophylaxis of Dysphagia After Radiotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kenneth Jensen, MD ph.d., University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20060059
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck cancer; Radiotherapy; Dysphagia; Exercise; Deglutition; Randomized controlled trial; Quality of life; Tube feeding
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Swallowing Exercises — Daily exercises

SUMMARY:
Background: Dysphagia is a common side effect after radiotherapy for haed and neck cancer patients. It may be worsened by immobility of the throat during tube feeding. Hypothesis: Exercises may prevent or reduce late dysphagia. Method: Phase I study to identify the tolerated intensity of exercises and establish the method of measuring training intensity and dysphagia measurement. Endpoint: Objective dysphagia using VF and FEESST. The HN swallowing and HN pain endpoint of EORTC H&N35 questionnaire. Weight loss, duration of tube feeding.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer
* Planned curative radiotherapy
* Planned irradiation of level II+III lymph nodes >46 Gy
* >=18 y
* Speaks and reads Danish
* No previous Surgery to the head and neck area except biopsies

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Objective swallowing using videofluoroscopy and endoscopic evaluation of swallowing | 2 mths

SECONDARY OUTCOMES:
Weight | 2 mths
Duration of tube feeding | 2 mths
Swallowing scale of EORTC HN 35 | 2 mths

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Jensen, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus, Denmark